CLINICAL TRIAL: NCT02415387
Title: The IMPACT Study: Inflammatory Responses, Mood and Physical Fitness After Cancer Treatment
Brief Title: Typhoid Vaccine in Testing Response to Immune Stress in Patients With Stage I-IIIA Breast Cancer
Acronym: IMPACT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OSU-13194; NCI-2014-01251 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Side Effects of Cancer Therapy; Depression; Recurrent Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Depression; Breast Neoplasms | interventions — Typhoid-Paratyphoid Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (inactive typhoid vaccine, placebo) (Experimental): Patients receive inactive typhoid vaccine IM at visit 1 followed by placebo IM 30 days later at visit 2.
  Interventions: Biological: typhoid vaccine; Other: Placebo
- Arm II (placebo, inactive typhoid vaccine) (Placebo Comparator): Patients receive placebo IM at visit 1 followed by inactive typhoid vaccine IM 30 days later at visit 2.
  Interventions: Biological: typhoid vaccine; Other: Placebo

INTERVENTIONS:
Biological: typhoid vaccine — Given IM
Other: Placebo — Given IM
  Other Names: PLCB

SUMMARY:
This randomized clinical trial uses an inactive typhoid vaccine to briefly stimulate an immune response in patients with stage I-IIIA breast cancer who received primary cancer treatment and studies whether patients' fitness levels affect how their bodies handle a challenge to their immune system. A vaccine is a substance or group of substances meant to cause the immune system to respond to a tumor or to microorganisms such as bacteria or viruses. Immune responses may cause excess inflammation in the body and behavioral changes, such as depression, fatigue, pain, and problems with thinking and reasoning. Studying immune responses in patients with breast cancer who have undergone primary cancer treatment may help doctors learn whether physical fitness can protect the body from effects of immune system stress and whether it may be able to reduce health problems in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the relationships between cardiorespiratory fitness and inflammatory and behavioral responses (negative mood, fatigue, pain, and cognitive problems) to typhoid vaccine in breast cancer survivors.

II. To determine the effects of age and depressive symptoms on inflammatory and behavioral responses to typhoid vaccine and placebo.

III. To assess the ability of cardiorespiratory fitness to moderate age- and depression-related responses to typhoid vaccine.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive inactive typhoid vaccine intramuscularly (IM) at visit 1 followed by placebo IM 30 days later at visit 2.

ARM II: Patients receive placebo IM at visit 1 followed by inactive typhoid vaccine IM 30 days later at visit 2.

There is an initial screening visit where patients in both arms complete an audio-recorded interview that includes questions about changes in mood and emotion throughout their lives, body measurements, a finger stick to assess for anemia and diabetes markers. During visit 1 and 2, patients in both arms will have blood drawn periodically and complete sets of questionnaires that assess feelings, health behaviors, and personality. Patients also complete cognitive tasks and a temperature sensitivity task at 3-4.5 hours post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been diagnosed with stage I-IIIA breast cancer will be recruited 1-10 years after the completion of all primary cancer treatment except for longer-term hormonal therapies (tamoxifen, aromatase inhibitors)
* All women will be postmenopausal

Exclusion Criteria:

* A prior history of any other malignancy except basal or squamous cell skin cancers, strokes, diabetes, current heart disease or uncontrolled hypertension, peripheral vascular disease, liver disease, autoimmune and/or inflammatory diseases including rheumatoid arthritis and ulcerative colitis, and other medical conditions that would limit participation in the assessments (e.g., pulmonary disease, orthopedic problems, major psychiatric illness, major cognitive dysfunction, or an acute medical problem)
* Anemia
* Alcohol or drug abuse
* Smoking
* Medication exclusions will include steroids as well as statins and other medications with anti-inflammatory actions
* Women who have received a typhoid vaccine within the last three years

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Kiecolt-Glaser, PhD, Principal Investigator — Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Wexner Medical Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madison AA, Renna M, Andridge R, Peng J, Shrout MR, Sheridan J, Lustberg M, Ramaswamy B, Wesolowski R, Williams NO, Noonan AM, Reinbolt RE, Stover DG, Cherian MA, Malarkey WB, Kiecolt-Glaser JK. Conflicts hurt: social stress predicts elevated pain and sadness after mild inflammatory increases. Pain. 2023 Sep 1;164(9):1985-1994. doi: 10.1097/j.pain.0000000000002894. Epub 2023 Mar 22. PMID 36943254
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Placebo/Vaccine): Patients receive placebo IM at visit 1 followed by inactive typhoid vaccine IM 30 days later at visit 2.
  typhoid vaccine: Given IM
  Placebo: Given IM
- Arm II (Vaccine/Placebo): Patients receive inactive typhoid vacccine IM at visit 1 followed by placebo IM 30 days later at visit 2.
  typhoid vaccine: Given IM
  Placebo: Given IM
Period: Overall Study
Arm/Group | Arm I (Placebo/Vaccine) | Arm II (Vaccine/Placebo)
Started | 87 | 85
Completed | 80 | 83
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 6 | 1
Not completed — blood draw problem | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Our 172 participants fell short of our 180 recruitment goal because COVID-19 issues.
Groups:
- All Participants: Patients served as her own control between two visits.
  typhoid vaccine: Given IM
  Placebo: Given IM
Arm/Group | All Participants
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 159
  More than one race | 2
  Unknown or Not Reported | 0
BMI [Count of Participants; unit: Participants]
  <18.5 kg/m^2 Underweight | 0
  18.5 kg/m^2 to 24.9 kg/m^2 Healthy | 61
  25 kg/m^2 to 29.9 kg/m^2 Overweight | 60
  >29.9 kg/m^2 Obese | 51
Trunk Fat [Mean (Standard Deviation); unit: kg] | 15.7 (6.7)
Vo2peak [Mean (Standard Deviation); unit: mL/kg/min] — Population: Peak oxygen consumption COVID-19 hospital protocols did not permit VO2 assessments on 14 women.
  mL/kg/min
    number analyzed (Participants) | 158
    (all) | 22.0 (5.3)
Years since treatment [Mean (Standard Deviation); unit: Years] | 3.5 (2.3)
Chemotherapy treatment [Count of Participants; unit: Participants] | 116
Radiation treatment [Count of Participants; unit: Participants] | 105
Cancer Stage [Count of Participants; unit: Participants]
  Stage I | 81
  Stage II | 82
  Stage III | 9
Comorbidities [Count of Participants; unit: Participants] | 22
CES-D score [Mean (Standard Deviation); unit: units on a scale] — Population: CES-D: Center for Epidemiological Studies-Depression. Scores range from 0 to 60, with higher scores indicating greater depressive symptoms.
  units on a scale | 7.5 (6.8)
Energy (SF-36 RAND) [Mean (Standard Deviation); unit: units on a scale] — Population: From SF-36 RAND Health Survey, scores range from 0 to 100, with higher scores indicating more energy or less fatigued.
  units on a scale | 60.4 (18.8)

OUTCOME MEASURES:

1. Primary Outcome: AUC Change in Level of IL-6
Description: AUC change refers to the 'net incremental' area, which is the area under the curve above the baseline value. Data points used in AUC change calculation include baseline, 1.5, 3, 5, 6.5, 8 hours post vaccine. This can be calculated geometrically by applying the trapezoid rule. When a value falls below the baseline, only the area above the baseline level is included.
Time Frame: Baseline, 1.5, 3, 5, 6.5, 8 hours post vaccine
Population: Each patient had two visits and served as her own control.
Measure: Least Squares Mean (Standard Error); unit: ug*hour/ml
Groups:
- Placebo: Placebo arm includes patients who got placebo injection no matter which sequence (vaccine/placebo or placebo/vaccine) was randomized into.
- Inactive Typhoid Vaccine: Inactive typhoid vaccine arm includes patients who got inactive typhoid vaccine injection no matter which sequence (vaccine/placebo or placebo/vaccine) was randomized into.
Arm/Group | Placebo | Inactive Typhoid Vaccine
Number analyzed (Participants) | 156 | 151
ug*hour/ml | 5.23 (0.27) | 10.17 (0.27)

2. Secondary Outcome: AUC Change in Pain
Description: Self-reported intensity of pain on 0-9 scale (0 = no pain; 9 = pain as bad as you can imagine). AUC change refers to the 'net incremental' area, which is the area under the curve above the baseline value. Data points used in AUC change calculation include baseline, 2, 3.5, 5, 6.5, 8.5 hours post vaccine. This can be calculated geometrically by applying the trapezoid rule. When a value falls below the baseline, only the area above the baseline level is included.
Time Frame: baseline, 2, 3.5, 5, 6.5, 8.5 hours post vaccine
Population: Each patient had two visits and served as her own control.
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hour
Arm/Group | Placebo | Inactive Typhoid Vaccine
Number analyzed (Participants) | 156 | 151
units on a scale*hour | 1.06 (0.50) | 3.24 (0.50)

3. Secondary Outcome: AUC Change in Fatigue
Description: Self-reported intensity of fatigue on 0-9 scales (0 = no fatigue; 9 = fatigue as bad as you can imagine). AUC change refers to the 'net incremental' area, which is the area under the curve above the baseline value. Data points used in AUC change calculation include baseline, 2, 3.5, 5, 6.5, 8.5 hours post vaccine. This can be calculated geometrically by applying the trapezoid rule. When a value falls below the baseline, only the area above the baseline level is included.
Time Frame: baseline, 2, 3.5, 5, 6.5, 8.5 hours post vaccine
Population: Each patient had two visits and served as her own control.
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hour
Arm/Group | Placebo | Inactive Typhoid Vaccine
Number analyzed (Participants) | 156 | 151
units on a scale*hour | 4.05 (0.77) | 3.62 (0.78)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Description: Any adverse events (AE) occurring during any part of the protocol will be reported immediately to the PI. A written report of all adverse events will be completed within 48 hours and submitted to the OSU IRB. Annually, IRB reports will include the occurrence of (un-) anticipated adverse events, and the timely progress of the trial, e.g. listing of all serious adverse events that occurred with clinical summaries, enrollment, withdraws, completions, etc.
Arm/Group | Placebo | Inactive Typhoid Vaccine
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/165
Other Adverse Events (participants affected / at risk) | 2/170 | 4/165
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=170) | Inactive Typhoid Vaccine (N=165)
Feeling ill (General disorders) | 2 (2) | 4 (4) — Headache, fatigue, nausea, dizzy, vomit, muscle pain

LIMITATIONS AND CAVEATS:
Our study focused on the initial, rapid inflammatory response, and we did not assess antibody responses to the vaccine, one limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02415387/Prot_SAP_000.pdf